CLINICAL TRIAL: NCT04048174
Title: Safety and Efficacy of Lactococcus Lactis Probiotic Bacteria for the Treatment of Chronic Rhinosinusitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: McGill University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CE12.288; 191920 (Other: Health Canada)
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-07

CONDITIONS: Chronic Rhinosinusitis
Keywords: Probiotics; Chronic rhinosinusitis; Irrigation; Microbiome

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline irrigation (Sham Comparator): Each participant performed nasal saline irrigation at 2 periods:
  * Day -14 to Day 0
  * Day 14 to Day 28
  Interventions: Other: Topical probiotic treatment with Lactococcus lactis W136; Other: Saline irrigation
- Probiotic lactococcus lactis W136 irrigation (Experimental): Each participant performed Probiotic lactococcus lactis W136 nasal irrigation from Day 0 to D14
  Interventions: Other: Topical probiotic treatment with Lactococcus lactis W136; Other: Saline irrigation

INTERVENTIONS:
Other: Topical probiotic treatment with Lactococcus lactis W136 — Nasal and sinus irrigation with reconstituted live probiotic bacteria
  Other Names: Natural health product
Other: Saline irrigation — Nasal and sinus irrigation with saline solution
  Other Names: Natural health product

SUMMARY:
Despite advances in medical treatments and surgery for chronic rhinosinusitis (CRS), there remains a large number of patients who continue to suffer from chronic sinusitis despite standard therapies. This research project has the goal of evaluating the safety and effectiveness of a potentially novel therapy for patients with CRS refractory to medical and surgical therapies, consisting of the introduction of a live probiotic bacteria (L lactis W136) directly into the nasal and sinus cavities via irrigation.

In total, 24 patients suffering from refractory CRS will be recruited from ongoing clinical activities by the research team of Martin Desrosiers at the CHUM hospital. Study duration is six weeks, and will be performed in three phases, with six visits planned in total.

1. Two-week observation period where only saline irrigation is administered.
2. Treatment period of 14 days (D0 to D14) during which L lactis W136 will be administered twice-daily.
3. Post treatment observation period of two weeks (D14 to D28) during which the patient will cease probiotic but will continue to irrigate his nose with only saline.

Assessment will use symptom questionnaires, quality of life questionnaires and endoscopic examination of the sinus cavities. Sinus culture will be performed at each visit to assess development of unusual infections. Exploratory assessments of gene expression and microbiome profiling will be performed to explore underlying mechanisms.

DETAILED DESCRIPTION:
CONTEXT/JUSTIFICATION:

Chronic rhinosinusitis (CRS) is one of the most frequent chronic diseases and has a significant negative impact on quality of life (QOL) in patients who suffer from it. Despite advances in medical treatments and surgery, there remains a large number of patients who continue to suffer from chronic sinusitis despite standard therapies. This research project has the goal of evaluating the safety and effectiveness of a potentially novel therapy for chronic sinusitis, via introduction of a probiotic bacteria (L lactis W136) directly into the nasal and sinus cavities via irrigation.

Probiotics are living micro-organisms (bacteria or fungi), which are added his compliments to certain dietary products such as yogurt to cereals with the intended effect of a beneficial effect on host health. The World Health Organization (WHO) and the league of the United Nations for Foodstuffs and Agriculture have defined probiotics as "living micro-organisms, which, when administered in sufficient quantity, exercise a positive effect on health beyond those of traditional nutritional benefits".

GOALS OF THERAPY:

To study the safety and clinical efficacy of an intranasal treatment with probiotic L lactis W136 in a population of patients with rhinosinusitis CRS refractory to medical and surgical therapies.

METHODOLOGY:

The study was performed in three phases, with six visits planned in total:

1. An observation period of two weeks (D-14 to D0) during which the patient will irrigate his/her sinuses only with saline solution. No other sinus medication will be allowed.
2. Treatment period of 14 days (D0 to D14) during which L lactis W136 will be administered twice daily in the form of 120 ml pf nasal irrigation solution containing dissolved probiotics in a buffered saline solution.
3. Surveillance Period: Post treatment observation period of two weeks (D14 to D28) during which the patient will cease probiotic but will continue to irrigate his nose with only saline solution and take no other sinus medication.

In order to assess the tolerance to treatment and the efficacy, selected patients will be examined at days D-14, D0, D1, D7, D14 and D28, and assessed according to a standardized scale. This assessment will be based on clinical criteria (sinus symptoms, quality-of-life assessments) endoscopic aspect of the mucosa and exploratory studies into molecular mechanisms of the microbiome and pathogenesis.

PREPARATION OF THE STUDY PRODUCT L Lactis is furnished by Agropur. Each patient will receive the probiotic in frozen individual doses. At time of use, these will be reconstituted into a 0.9% solution. This will be administered to the nose via nasal irrigation using the NeilMed Paediatric Sinus Rinse apparatus which contains 120 cc.

STUDY TREATMENT Nasal irrigation with 1.2 x 10e9 CFU of L. Lactis dissolved in 120mL of 0.9% saline solution administered BID to both nostrils for 14 days.

Recruitment of study participants

Patients will be recruited form ongoing clinical activities. Recruitment will be by a staff member not associated with clinical care. After explanation of the study and informed consent, patients will have a complete ENT history and examination including nasal endoscopy to confirm admissibility.

In addition, the patient will complete questionnaires on sino nasal symptoms and a sinus-specific quality of life (SNOT-22)

Pregnancy tests will be performed on all female participants of reproductive potential.

CRITERIA FOR EARLY WITHDRAWAL / PREMATURE TERMINATION

* Incapable of performing nasal irrigation
* Severe irritation of the nose and sinus mucosa
* Signs and/or symptoms of acute infection
* Development of otitis (ear infection)

Antidote Oral antibiotic

Washout period There will be a washout period of fourteen days prior to probiotic administration during which the only permitted sinus medication will be continued use sinus irrigation.

Concomitant Medication No rescue medication is planned for in this study.

Clinical parameters assessed :

1. Clinical criteria Total nasal and sinus symptoms (0-3 scale) Disease specific Quality of life (QOL) SNOT-22 Surveillance of adverse effects
2. Endoscopic criteria Direct examination of the sinus mucosa using a 0-degree endoscope. Grading according to the POSE system.
3. Markers of inflammation Mucosal brushings will be obtained at the level of the frontal recess using a cytology brush. RNA will be extracted and processed for gene expression profiling to explore underlying mechanisms.
4. Composition of the microbiome Conventional sinus cultures will be performed at each visit to monitor infection / probiotic overgrowth. Microbiome profiling will be performed using 16S sequencing on swabs taken form the sinuses.

EFFICACY ANALYIS

* Sino-nasal symptomatology and quality of life indices
* Direct endoscopic assessment of the sinus mucosa

Safety Analyses

* Tolerability of L lactis intranasally will be assessed on Day by questionnaire, examination and nasal endoscopy.
* Potential impact on adjacent structures :
* Olfactive zone of the nose will be assessed by UPSIT smell tests Eustachian tube: Middle ear examination with microscopy

Statistical Analysis At days -14, 0, 7, 14 and 28 after treatment, subjective and endoscopic results will be analysed using Brapkar's test for paired qualitative observations.

ELIGIBILITY:
Inclusion Criteria:

* refractory chronic rhinosinusitis (CRS)
* persistence of symptoms of CRS despite previous endoscopic sinus surgery (ESS) and ongoing medical management

Exclusion Criteria:

* patients <18 years
* cystic fibrosis
* technical reasons for ESS failure
* active sinus infection with purulence pain and/or hyperthermia
* immune suppression from disease or medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-03-06 (Actual); Primary Completion 2015-12-02 (Actual); Study Completion 2015-12-02 (Actual)

PRIMARY OUTCOMES:
Sino-nasal symptom score | 6 weeks
  Subjective symptoms of nasal function.
  The sino-nasal symtom score (SNSS) is the sum of the following nasal and sinus symptoms:
  1. Nasal obstruction
  2. Facial pain
  3. Need to blow nose
  4. Headache
  5. Post-nasal drip
  Each individual item is scored on a 0-3 ordinal scale, with a higher score indicating a worst/more severe symptom. The TNSS is the sum of the five symptoms and has a range of 0-15. A lower score is better.

SECONDARY OUTCOMES:
SNOT-22 | 6 weeks
  SNOT-22 validated disease - specific quality of life score. The Sino-Nasal Outcome Test is a validated, disease specific quality of life questionnaire. It contains 22 items, which contributes to the SNOT-22 acronym. Each of the individual items is scored on a 0-5 ordinal score. A higher score indicate worst quality of life. Individual results are summed with equal weight. The sum is the SNOT-22 score, which has a range of 0-110. A lower score is better.
Post Operative Sinus Endoscopy Score (POSE) | 6 weeks
  Validated endoscopic scoring system. The Perioperative Sinus Endoscopy score assesses the condition of the sinuses and sinus mucosa as assessed with direct endoscopic visualization of the sinus passages. Presence of oedema, polyps, scarring and nasal secretions, and status of the principal sinus drainage passages (frontal and sphenoid), are assessed on a 0-2 ordinal scale. A higher score indicate worse disease.
  POSE score is determined as the sum of each of the individual items and has a range of 0-12.
Sinus culture (conventional) | 6 weeks
  Swab culture for monitoring of infection/probiotic over growth

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Endam LM, Alromaih S, Gonzalez E, Madrenas J, Cousineau B, Renteria AE, Desrosiers M. Intranasal Application of Lactococcus lactis W136 Is Safe in Chronic Rhinosinusitis Patients With Previous Sinus Surgery. Front Cell Infect Microbiol. 2020 Oct 12;10:440. doi: 10.3389/fcimb.2020.00440. eCollection 2020. PMID 33154953